CLINICAL TRIAL: NCT06830590
Title: Study of Molecular Characterisation of Early Operable Primary Breast Cancer in Pakistani Population
Acronym: BrCa
Status: Recruiting | Type: Observational
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Prof. Binafsha Manzoor Syed, Prof. Dr., Liaquat University of Medical & Health Sciences
Other Study IDs: BreastCa001
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Molecular Pathway Deregulation; Treatment
Keywords: Breast cancer; Molecular characterisation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — FFPE blocks of breast tumors will be retained
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early operable primary breast cancer: 1. women
  2. any age group
  3. confirmed diagnosis of breast cancer
  Interventions: Procedure: Molecular characterisation

INTERVENTIONS:
Procedure: Molecular characterisation — All patients treated by surgery were included without any neoadjuvant therapy

SUMMARY:
This study is looking at the biological characteristics of early operable primary breast cancer in Pakistani Population by using IHC

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed diagnosis of breast cancer without history of taking neoadjuvant therapy Good quality tumour samples available for IHC

Exclusion Criteria:

* patients received pre-operative chemotherapy or radiotherapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Females only
Study Population: The population are women with early operable primary breast cancer underwent surgery without any prior treatment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Breast cancer specific survival in correlation with molecular pattern | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Binafsha Manzoor M Syed, MBBS, PhD, Principal Investigator — Liaquat University of Medical & Health Sciences, Jamshoro
Locations (1):
- Binafsha M Syed, Jamshoro, Pakistan

IPD SHARING:
Plan to Share IPD: No
data will be shared in the form of overall results with pattern of biomarkers. Individual participants data will not be shared